CLINICAL TRIAL: NCT00403442
Title: Bevacizumab in Combination With Verteporfin Reduced and Standard Fluence in the Treatment of Hemorrhaged Lesions in Neovascular AMD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: QLT Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2303
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Device: Verteporfin Therapy/ Drug: Bevacizumab

SUMMARY:
The purpose of this study is to explore the combination of PDT with verteporfin at reduced and standard fluence rates, in conjunction with bevacizumab, in the treatment of subfoveal CNV of all subtypes with a high percentage of subretinal hemorrhage (hemorrhage >50% of total lesion area).

To assess the safety of bevacizumab in combination with verteporfin PDT (reduced fluence: 300 mW/cm2) as compared to bevacizumab in combination with verteporfin PDT (standard fluence: 600 mW/cm2) in patients whose neovascular CNV lesions containing >50% blood.

DETAILED DESCRIPTION:
This is a phase one study in patients with all CNV lesion subtypes who are naïve to previous treatment. Lesions must have blood as a primary component (i.e., contain more than 50% blood). Patients will receive one of two combination treatments:

* Verteporfin PDT reduced fluence (300 mW/cm2) immediately followed by bevacizumab (1.25 mg) intravitreal injection
* Verteporfin PDT standard fluence (600 mW/cm2) immediately followed by bevacizumab (1.25 mg) intravitreal injection A total of 10 patients will be enrolled, 5 per treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients are men or women of age 50 or older.
* Patients diagnosed with subfoveal CNV due to AMD with lesion size ≤6 DA.
* Patients have not received previous treatment for subfoveal CNV, in the study eye.
* Patients with visual acuities at baseline between 20/40 and 20/320, as evaluated on ETDRS scale.
* Fluorescein Angiography showing any type of subfoveal CNV at baseline with >50% blood component of total lesion area.

Exclusion Criteria:

* Patients with a known hypersensitivity/allergy to verteporfin, porfimer sodium, or other porphyrins, porphyria or other porphyrin sensitivity, or hypersensitivity to sunlight or bright artificial light.
* Patients with history of glaucoma requiring treatment, or are currently on antihypertensive treatment for elevated intraocular pressure.
* Women of childbearing potential must not be pregnant of lactating, must have a negative pregnancy test at screening and must be practicing an adequate method of birth control.
* Patients who have had treatment for CNV in the study eye with photodynamic therapy (PDT), transpupillary thermotherapy (TTT), or other local treatment (e.g. submacular surgery, intravitreal triamcinolone, intra-ocular antiangiogenic agents). Previous laser photocoagulation therapy is acceptable, provided it was not subfoveal.
* Subject's currently who have been involved in any experimental procedure within the last 12 weeks.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
The primary safety variable is visual acuity and adverse events at Month 12.

SECONDARY OUTCOMES:
Change in percentage of lesion hemorrhage from baseline.
The proportion of patients who lose fewer than 15 letters Less than 3 lines of best corrected visual acuity in the study eye from baseline
The proportion of patients who gain 15 letters or more greater or equal to 3 lines of best-corrected visual acuity in the study eye from baseline
Mean change from baseline in best-corrected visual acuity score. OCT evidence of active CNV leakage which may include persistent retinal edema, subretinal
fluid or pigment epithelial detachment. FA evidence of active CNV leakage which may include subretinal fluid or hemorrhage.
Number of retreatments, bevacizumab and verteporfin PDT, at either fluence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Slakter, M.D., Principal Investigator — Vitreous Retina Macula Consultants of New York, P.C.
Locations (1):
- Vitreous Retina Macula Consultants of New York, P.C., New York, New York, United States